CLINICAL TRIAL: NCT04119570
Title: Pilot and Trial of the Chronic Kidney Disease Report Card
Brief Title: CKD Report Card Pilot Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-0283
Record Dates: First submitted 2019-09-17; First posted 2019-10-08 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: CKD

STUDY DESIGN:
Intervention Model Description: During the first half of the study, participants will be surveyed and observed without the intervention. During the second half, participants will be surveyed and observed with the intervention (CKD Report Card)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intervention (No Intervention): Participants will have their clinic visit as per usual care.
- CKD Report Card (Active Comparator): Participants will receive the CKD Report Card prior to the clinic visit.
  Interventions: Behavioral: CKD Report Card

INTERVENTIONS:
Behavioral: CKD Report Card — The CKD Report Card is a handout based on a NKDEP Educational Sheet that includes basic information about kidney disease and spaces where patient can record information about their own kidney disease
  Arms: CKD Report Card

SUMMARY:
The investigators will study physician-patient communication at the UCMC nephrology fellow clinic and to test an intervention, the CKD Report Card, to improve that communication and patient knowledge of CKD.

DETAILED DESCRIPTION:
The goals of the study are to 1) characterize the effectiveness and patient-centeredness of patient-physician interaction during a nephrology clinic visit both with and without use of the CKD Report Card, and 2) to determine which physician and patient characteristics are associated with effective and patient centered communication. There will be block enrollment. For Nephrology physicians who agreed to participate will complete a baseline questionnaire. Research assistants will approach patients of participating providers in clinic waiting rooms, with the goal of enrolling patients for each provider For half of the study, investigators will enroll patients in the study and observe patient-physician communication and use a survey measure CKD knowledge pre-visit and post-visit. For the second half of the study, investigators will give participants the CKD Report Card, an investigator-developed handout, to use during the clinic visit. Investigators will observe patient-physician communication and use a survey to measure CKD knowledge pre-visit and post-visit. For both groups, eligible participants will give informed consent and will complete a baseline questionnaire; research assistants will place a digital audio-recording device in the examination room to record the patient-provider encounter. Following the medical encounter, research assistants will administered an interview with patients, assessing demographic, social, and behavioral characteristics, as well as their experience of care and ratings of provider communication.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking adult patients (age 18 or older)
* Identified in the medical record as non-Hispanic Black or non- Hispanic White
* seen in University of Chicago nephrology clinic with a participating nephrologist

Exclusion Criteria:

* not able to communicate in English
* lacking ability to consent to study
* does not identify as non-Hispanic Black or non-Hispanic
* without chronic kidney disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
CKD Knowledge | Change in CKD Knowledge from Baseline (pre-visit) to CKD Knowledge immediately post clinic visit (within 15-100 minutes post-clinic visit)
  Kidney Disease Knowledge Survey (KiKs)

SECONDARY OUTCOMES:
patient-physician interaction | immediately post-nephrology clinic visit (on day of enrollment, within 15-100 minutes post-clinic visit)
  Perceived efficacy in patient-physician interactions (PEPPI)
communication assessment | immediately post-nephrology clinic visit (on day of enrollment, within 15-100 minutes post-clinic visit)
  communication assessment tool (CAT)

CONTACTS AND LOCATIONS:
Overall Officials: Milda R. Saunders, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No